CLINICAL TRIAL: NCT03356574
Title: Long-term Survival After Single-ventricle Palliation: A Swedish Nationwide Cohort Study
Brief Title: Long-term Survival After Single-ventricle Palliation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Queen Silvia Children's Hospital, Gothenburg, Sweden (Other); Lund University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, PhD, Principal Investigator, Karolinska University Hospital
Other Study IDs: Single-ventricle survival
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Single-ventricle palliation surgery — Single-ventricle palliation surgery

SUMMARY:
A nationwide observational study. Children operated with single-ventricle palliation between January 1994 and December 2017 operated in Sweden will be included retrospectively. Patients born with a functionally single ventricle but not undergoing surgery will not be included. Data regarding preoperative clinical characteristics and operative details will be obtained by medical records review and from The Swedish Registry of Congenital Heart Disease (SWEDCON). Using unique personal identity numbers assigned to all residents of Sweden, data from SWEDCON will be linked with dates of death.

ELIGIBILITY:
Inclusion Criteria:

* Operated with single-ventricle palliation between January 1994 and May 2017 in Sweden.

Exclusion Criteria:

* None.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children operated with single-ventricle palliation between January 1994 and May 2017 in Sweden.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1994-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | Until death or end of follow-up (December 31st 2017)

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Pediatric Heart Center, Queen Silvia Children's Hospital, Gothenburg
  - Pediatric Heart Center, Lund University Hospital, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalen M, Odermarsky M, Liuba P, Johansson Ramgren J, Synnergren M, Sunnegardh J. Long-Term Survival After Single-Ventricle Palliation: A Swedish Nationwide Cohort Study. J Am Heart Assoc. 2024 Mar 19;13(6):e031722. doi: 10.1161/JAHA.123.031722. Epub 2024 Mar 18. PMID 38497454